CLINICAL TRIAL: NCT00217516
Title: Supplementation of L-Selenomethionine in Patients With Prostate Cancer Prior to Brachytherapy. Selenium Brachytherapy Trial: Phase I/Pilot Study
Brief Title: Selenium in Treating Patients Who Are Undergoing Brachytherapy for Stage I or Stage II Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000441225; P30CA016056 (NIH); RPCI-I-14603
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2012-02-09 (Estimated); Status verified 2010-09

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage I prostate cancer; stage II prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Selenium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients receive oral selenium for 3-6 weeks.
  Interventions: Drug: selenium
- Arm II (Placebo Comparator): Patients receive oral placebo for 3-6 weeks.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: selenium — Given orally
  Arms: Arm I
Other: placebo — Given orally
  Arms: Arm II

SUMMARY:
RATIONALE: The use of nutritional supplements, such as selenium, may stop prostate cancer from growing. Internal radiation, such as brachytherapy, uses radioactive material placed directly into or near a tumor to kill tumor cells. Giving selenium before brachytherapy may be an effective treatment for prostate cancer.

PURPOSE: This randomized phase I trial is studying selenium to see how well it works compared to placebo in treating patients who are undergoing brachytherapy for stage I or stage II prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the effects of selenium vs placebo on tissue biomarkers of prostate cancer susceptibility, using tissue samples from biopsies before and after treatment, in patients undergoing brachytherapy for stage I or II prostate cancer.

Secondary

* Determine the effects of selenium on antioxidant enzyme activities in these patients.
* Determine, preliminarily, whether there is a threshold effect among patients with low baseline levels of selenium treated with this drug.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral selenium for 3-6 weeks. Patients then undergo brachytherapy.
* Arm II: Patients receive oral placebo for 3-6 weeks. Patients then undergo brachytherapy.

After completion of study treatment, patients are followed at 1 and 6 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate

  * Must have undergone ≥ a sextant biopsy
  * Clinical stage T1a-T2a disease
* Gleason score < 8
* Prostate-specific antigen < 20 ng/mL

PATIENT CHARACTERISTICS:

Age

* Not specified

Performance status

* Not specified

Life expectancy

* More than 5 years

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* No other prior malignancy except nonmelanoma skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* No prior hormonal therapy

Radiotherapy

* No prior radiotherapy

Surgery

* Not specified

Other

* More than 30 days since prior and no concurrent participation in another clinical trial involving a medical, surgical, nutritional, or lifestyle intervention (e.g., dietary modification or exercise)
* No selenium at doses > 50 mcg/day as a dietary supplement, including multivitamin supplements

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2005-03; Primary Completion 2008-02 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Effects of selenium vs placebo on tissue biomarkers of prostate cancer susceptibility at 1 and 6 months after completion of study treatment | 1 and 6 months after completion of study treatment

SECONDARY OUTCOMES:
Effects of selenium on antioxidant enzyme activities at 1 and 6 months after completion of study treatment | 1 and 6 months after completion of study treatment
Threshold effect among patients with low baseline levels of selenium at 1 and 6 months after completion of study treatment | 1 and 6 months after completion of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Michael R. Kuettel, MD, PhD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States